CLINICAL TRIAL: NCT06409026
Title: Effect of Sotatercept on Central Cardiopulmonary Performance and Peripheral Oxygen Transport During Exercise in Pulmonary Arterial Hypertension
Brief Title: Sotatercept on Central Cardiopulmonary Performance and Peripheral Oxygen Transport During Exercise in Pulmonary Arterial Hypertension
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Yogesh Reddy, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-002570
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ACE-011

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sotatercept Therapy (Experimental): All participants will receive 36 weeks of sotatercept therapy. Sotatercept is administered as a subcutaneous injection once every 3 weeks.
  Interventions: Drug: Sotatercept

INTERVENTIONS:
Drug: Sotatercept — As per FDA indications, sotatercept will be administered as 0.3 mg/kg injection for the first dose followed by 0.7 mg/kg injections for subsequent doses.

SUMMARY:
The purpose of this study is to see if the drug sotatercept given for 36 weeks improves the functioning of the heart and improves quality of life.

ELIGIBILITY:
Inclusion Criteria

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
* NYHA Class II-IV.
* LVEF ≥ 40 % within the preceding year.
* No recent initiation of pulmonary vasodilator in the last 60 days.
* Pulmonary arterial hypertension by right heart catheterization (Mean PA pressure ≥ 20 mmHg with PVR>2 Wood units) with no evidence of heart failure with preserved ejection fraction (exercise PCWP <25 mm Hg).
* Symptomatic PAH patients with plan to undergo exercise RHC for reassessment of exertional symptoms.

Exclusion Criteria

* Myocardial infarction, stroke, hospitalization for heart failure, unstable angina pectoris or transient ischemic attack within 30 days prior to the day of screening.
* Planned coronary, carotid, or peripheral artery revascularization.
* Any other condition judged by the investigator to be the primary cause of dyspnea (such as heart failure due to restrictive cardiomyopathy or infiltrative conditions (e.g., amyloidosis), hypertrophic obstructive cardiomyopathy, anemia, or more than moderate mitral or aortic heart valve disease).
* Wheelchair bound or orthopedic inability to exercise.
* Chronic hypoxemia with inability to exercise without oxygen supplementation.
* Skeletal muscle myopathy.
* History of rhabdomyolysis.
* Participation in any clinical trial of an approved or non-approved device for the treatment of pulmonary hypertension within 30 days before screening.
* Receipt of any investigational medicinal product within 30 days before screening.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method.
* Major surgery scheduled for the duration of the trial, affecting walking ability in the opinion of the investigator.
* Any disorder, including severe psychiatric disorder, suicidal behavior within 90 days before screening, and suspected drug abuse, which in the investigator´s opinion might jeopardize subject´s safety or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-05 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Pulmonary arterial mean pressure/Cardiac Output (PA/CO) at peak exercise | Baseline, Week 24
  Peak exercise pulmonary arterial mean pressure/ Cardiac output (mm Hg/L/min)

SECONDARY OUTCOMES:
Oxygen Consumption (VO2) | Baseline, 24 weeks
  VO2 will be measured in mL/kg/min. It will be directly measured using expired gas analysis.
Single leg blood flow at peak exercise | Baseline, 24 weeks
  Single leg blood flow will be obtained from venous access. Single leg blood flow will be measured in ml/min
Pulmonary vascular resistance at rest | Baseline, 24 weeks
  Pulmonary vascular resistance will be measured in Wood units (mmHg/L/min)
Pulmonary vascular resistance at peak exercise | Baseline, 24 weeks
  Pulmonary vascular resistance will be measured in Wood units (mmHg/L/min)
Pulmonary arterial (PA) compliance at rest | Baseline, 24 weeks
  PA compliance measures pulmonary arterial distensibility and will be recorded at Baseline and 24 Weeks. PA compliance will be measured in ml/mm Hg.
Pulmonary arterial (PA) compliance at peak exercise | Baseline, 24 weeks
  PA compliance measures pulmonary arterial distensibility and will be recorded at Baseline and 24 Weeks. PA compliance will be measured in ml/mm Hg.
Pulmonary arterial elastance at rest | Baseline, 24 weeks
  PA elastance measures pulmonary artery stiffness and will be recorded at baseline and 24 weeks as PA systolic pressure/stroke volume (units mm Hg/ml)
Pulmonary arterial elastance at peak exercise | Baseline, 24 weeks
  PA elastance measures pulmonary artery stiffness and will be recorded at baseline and 24 weeks as PA systolic pressure/stroke volume (units mm Hg/ml)
Left ventricular (LV) transmural pressure at rest | Baseline, 24 weeks
  LV transmural pressure will measured by catheterization at Baseline and 24 Weeks as the difference between pulmonary capillary wedge pressure and right atrial pressure
Left ventricular (LV) transmural pressure at peak exercise | Baseline, 24 weeks
  LV transmural pressure will measured by catheterization at Baseline and 24 Weeks as the difference between pulmonary capillary wedge pressure and right atrial pressure
Right Ventricular Pulmonary Artery Coupling at rest | Baseline, 24 weeks
  Calculated as the ratio of RV function by echocardiography indexed to PA systolic pressure (unit mmHg-1)
Right Ventricular Pulmonary Artery Coupling at peak exercise | Baseline, 24 weeks
  Calculated as the ratio of RV function by echocardiography indexed to PA systolic pressure (unit mmHg-1)
Eccentricity index at rest | Baseline, 24 weeks
  Eccentricity index will be calculated as the ratio of antero posterior and septolateral dimension of the left ventricle by echocardiogram
Eccentricity index at peak exercise | Baseline, 24 weeks
  Eccentricity index will be calculated as the ratio of antero posterior and septolateral dimension of the left ventricle by echocardiogram
Right atrial pressure (RA) at rest | Baseline, 24 weeks
  RA pressure (mm Hg) will be measured by catheterization conducted at Baseline and 24 weeks
Right atrial pressure (RA) at peak exercise | Baseline, 24 weeks
  RA pressure (mm Hg) will be measured by catheterization conducted at Baseline and 24 weeks
Change in skeletal muscle O2 diffusive conductance (Dm) during peak exercise | Baseline, 24 weeks
  Dm is measured in ml/mm Hg/min during peak exercise
Change in skeletal muscle O2 diffusive conductance (Dm) during single leg exercise | Baseline, 24 weeks
  Dm is measured in ml/mm Hg/min during single leg exercise

CONTACTS AND LOCATIONS:
Overall Officials: Yogesh Reddy, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No